CLINICAL TRIAL: NCT03059524
Title: Dynamic Monitoring of Circulating microRNA Changes in Patients With or Without Multiple Organ Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: Chengdu Nuoen Biotechnologies, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Uestc501
Record Dates: First submitted 2017-01-09; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Multiple Organ Failure
Keywords: microRNA
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood extraction from subjects subsequently separated to plasma.

GROUPS / COHORTS (3):
- patients with multiple organ failure
- patients without multiple organ failure
- normal subjects

SUMMARY:
The objectives are to:

1. validate a panel of tissue-specific miRNAs that are differentially expressed in the plasma of patients with and without multiple organ failure.
2. investigate the dysregulation of circulating miRNA panel and their prognostic and predictive values in clinical outcomes in identifying patients at high risk for mortality and multiple organ failure.

This trial involves peripheral blood sampling from subjects at their earliest presentation and remaining stays in the hospitalization in the emergency department. The investigators will develop panels of miRNAs that are specific indicator of early onset of major organ failures, and correlate clinical outcomes with these miRNAs.

DETAILED DESCRIPTION:
The ICU patients with multiple organ failure in sponsor's institutes will be enrolled in this observational cohort of investigation. Whole blood samples will be separated immediately into plasma for storage. The participants will have their 2nd and 3rd samples obtained at 24-48 hours and 48-72 hours respectively. The schedule of most of sampling schedule is designed in concordance with the ICU routines to avoid extra burdens on patients. The plasma samples will be used as prognostic markers in prognostic and predictive values in identifying patients at high risk for mortality and multiple organ failure. Patients who are discharged will be tracked for any clinical recurrence of the diseases every 28 days to assess the diagnostic accuracy of the miRNA biomarkers that are measured.

The 2nd objective will be assessed by measuring the concentration of miRNAs in normal patients without multiple organ failure.

The circulating miRNAs will be detected directly from 1 - 5 ul of plasma samples with the miRFLP assay. This capillary electrophoresis-based miRNA quantification method detects multiple miRNAs in absolute copy number in smaller sample signature with negligible batch to batch variation, thus providing a standard miRNA detection method.

ELIGIBILITY:
Inclusion Criteria for subjects:

* Adults 18 years and above
* Has condition related to ICU enrollment cause

Exclusion Criteria for subjects:

* Age below 18 years
* Known pregnancy
* Treating physician deems aggressive care unsuitable
* Unable to provide informed consent or comply with study requirements

Inclusion criteria for normal controls:

• Adults 18 years and above

Exclusion criteria for normal controls:

* Underlying chronic inflammatory condition (e.g. inflammatory bowel disease)
* Underlying autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus)
* Pre-existent liver disorder
* User of any prescript medicine or over the counter drugs in prior 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research project will recruit a cohort of prospective observational cancer patients in ICU. Admitted patients will be followed-up in the inpatient units in concordance with ICU protocols. Upon discharged, patients will be followed-up in every 28 days for any disease recurrence and clinical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The concentration of circulating miRNA expression quantitated in absolute copy numbers in ICU patients with or without multiple organ failures. | 3 years
  The circulating miRNA concentration is to be measured in patient plasma samples with or without multiple organ failures. The comparison of miRNA expression will be performed to investigate the potential prognostic value of the miRNA panel on survival rates at the onset of multiple organ failures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China